CLINICAL TRIAL: NCT03324048
Title: A Single Mindfulness Meditation Session in Preoperative Anxiety : Effects on the Autonomous Nervous System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 1708097; ID-RCB (Other: 2017-A01727-46)
Record Dates: First submitted 2017-10-05; First posted 2017-10-27 (Actual); Last update posted 2019-05-17 (Actual); Status verified 2018-07

CONDITIONS: Anxiety; Relaxation
Keywords: Preoperative anxiety; Relaxation; Autonomous nervous system; Surgery; Visual Analogue Scale (VAS); State-Trait Anxiety Inventory (STAI-Y)
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients anxious (Other): Patients anxious will be perform relaxation session.
  Interventions: Other: relaxation session

INTERVENTIONS:
Other: relaxation session — During relaxation session, patients anxious will have three electrodes for save heart rate variability and a sensor for save value of the partial pressure of carbon dioxide.
  Before and after relaxation session, patient evaluates his anxiety by visual analogue scale (VAS) and State-Trait Anxiety Inventory (STAI-Y).

SUMMARY:
Anxiety is an emotional disorder. It's a painful concern caused by uncertainty. It is a complex phenomenon misunderstood in spite of medical progress. Relaxation is a technical for reduce anxiety and is effective and safe. Previous study demonstrated the impact of session relaxation on the autonomous nervous system by the heart rate variability.

Primary objective of this new study is to demonstrate a link between heart rate variability and reduced anxiety during relaxation session.

DETAILED DESCRIPTION:
It is monocentric, prospective and interventional study. This study will be proposed at the patients who will have an orthopedic surgery in full hospitalization. These patients are anxious because of surgery too. The day before surgery anesthetist save heart rate variability and value of the partial pressure of carbon dioxide during relaxation session.

ELIGIBILITY:
Inclusion Criteria:

* Affiliated or entitled to a social security
* Have signed consent before their participation in the study
* Aged over 18 years
* Patients who will have an orthopedic surgery in full hospitalization
* Patients anxious on visual analogic scale of anxiety (>5)

Exclusion Criteria:

* Different disorder : disability to understand instructions, respiratory insufficiency, obesity, sleep apnea, wearing a pacemaker
* Medical history of schizophrenia or bipolar disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2017-11-14 (Actual); Primary Completion 2018-09-17 (Actual); Study Completion 2018-09-17 (Actual)

PRIMARY OUTCOMES:
high frequency | continuously during the relaxation session
  from the variation of heart rate. Measured by electrocardiogram.

SECONDARY OUTCOMES:
anxiety | after the relaxation session at day 1
  Measured with the State-Trait Anxiety Inventory (STAI-Y) Interpretation : Very high:> to 65 High: from 56 to 65 Average: from 46 to 55 Low: from 36 to 45 Very low: <or = 35
low frequency | continuously during the relaxation session
  Measured by electrocardiogram.
the ratio of high frequencies to low frequencies | continuously during the relaxation session
  Measured by electrocardiogram.
PetCO2 | continuously during the relaxation session
  measured with a sensor fixed in front of the nostril

CONTACTS AND LOCATIONS:
Overall Officials: Zeina PRADES, MD PhD, Principal Investigator — CHU SAINT-ETIENNE
Locations (1):
- CHU de SAINT-ETIENNE, Saint-Etienne, France

IPD SHARING:
Plan to Share IPD: No